CLINICAL TRIAL: NCT06880952
Title: Effect of Post-operative Chlorhexidine on Postoperative Pain and Complications After Surgical Removal of Mandibular Third Molars: a Randomized Controlled Trial
Brief Title: Effect of Post-operative Chlorhexidine on Postoperative Pain and Complications After Surgical Removal of Mandibular Third Molars
Acronym: RITOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jeroen van der Sleen, Oral Surgeon and Principal Investigator, Isala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 71727.075.20
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Third Molars Extraction
Keywords: third molar; chlorhexidine
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-operative rinsing with chlorhexidine (Other): In the rinsing group, the patients received a bottle of 0,2% chlorhexidine
  Interventions: Other: Chlorhexidine Digluconate Mouthwash without Alcohol
- No post-operative rinsing (No Intervention): Those allocated to the control group received no post-operative rinsing

INTERVENTIONS:
Other: Chlorhexidine Digluconate Mouthwash without Alcohol — In the rinsing group, the patients received a bottle of 0,2% chlorhexidine
  Arms: Post-operative rinsing with chlorhexidine

SUMMARY:
This study aimed to assess the impact of postoperative chlorhexidine use on pain management following mandibular third molar removal

In this prospective, randomized controlled trial,130 patients who underwent mandibular third molar surgical removal were divided into two groups: one group used chlorhexidine for postoperative rinsing and the other did not rinse. Pain levels, measured using the Numeric Rating Scale (NRS), were recorded daily for the first seven days post-surgery. Paired-samples t-tests were utilized for data analysis.

ELIGIBILITY:
Inclusion Criteria:

• healthy adults (18+) referred by their dentist for third molar removal

Exclusion Criteria:

* active pericoronitis or other infections
* planned coronectomy
* trismus
* chronic pain
* pregnancy
* known allergies to local anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Postoperative pain after removal of third molar | 7 days after the inclusion pain was measured on a numerical rating scale
  The primary endpoint is the difference in the postoperative pain measured on a numerical rating scale (NRS) evaluated at seven days

SECONDARY OUTCOMES:
Post-operative complications | 7 days after the treatment the patient was seen at the outpatient clinic for clinical assessment. At this moment the number of patients with alveolitis, foodimpaction and bleeding was scored.
  As secondary outcome measures alveolitis, foodimpaction, bleeding or infection

CONTACTS AND LOCATIONS:
Locations (1):
- Isala Hospital, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghaeminia H, Hoppenreijs TJ, Xi T, Fennis JP, Maal TJ, Berge SJ, Meijer GJ. Postoperative socket irrigation with drinking tap water reduces the risk of inflammatory complications following surgical removal of third molars: a multicenter randomized trial. Clin Oral Investig. 2017 Jan;21(1):71-83. doi: 10.1007/s00784-016-1751-1. Epub 2016 Feb 27. PMID 26922634